CLINICAL TRIAL: NCT01940653
Title: Optimal Length of Progesterone Supplementation Before the Transfer of Cryopreserved (Frozen)-Thawed Day 3 Embryos in an Artificial Cycle With Exogenous Estrogen and Progesterone
Acronym: PROFETA-3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Arne van de Vijver, Medical Doctor, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROFETA-3
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Progesterone Supplementation
MeSH Terms: interventions — Progesterone; Estradiol; Utrogestan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Progesterone (Other): Group A receives 5 days of micronized progesterone vaginally (Utrogestan® ((Utrogestan, Besins International). On the 5th (group A) of progesterone supplementation, the cryopreserved-thawed day 3 embryo is transferred.
  Interventions: Drug: Progesterone
- progesterone 3 days (Active Comparator): Group B receives 3 days of micronized progesterone vaginally. On the 3rd day of progesterone supplementation, the cryopreserved-thawed day 3 embryo is transferred.
  Interventions: Drug: Progesterone

INTERVENTIONS:
Drug: Progesterone — Procedures Transvaginal ultrasound (US) and hormone analysis for FSH, LH, E2 and P on day 2 of the cycle will be performed. The artificial preparation of the endometrium consists of 7 days oestradiol valerate (Progynova®, Bayer-Schering Pharma AG, Berlin, Germany) 2 mg bid (bi-daily), followed by 6 days oestradiol valerate 2 mg tid (thrice daily). On day 13, the endometrium is measured. If endometrial thickness is more than 7 mm, patients are randomly assigned to group A or B. All patients with an endometrium less than 7 mm on day 13 of estrogen stimulation, are excluded.
  Group A receives 5 days of micronized progesterone vaginally (Utrogestan® ((Utrogestan, Besins International), 3x200mg daily), group B receives 3 days of micronized progesterone vaginally. On the 5th (group A) or 3rd (group B) day of progesterone supplementation, the cryopreserved-thawed day 3 embryo is transferred.
  Other Names: oestradiol valerate (Progynova®, Bayer-Schering Pharma AG, Berlin, Germany); progesterone (Utrogestan®, Besins International, France)

SUMMARY:
Cryopreserved-thawed embryos are often replaced in an artificial cycle, in which the endometrium is prepared by exogenous estrogen and progesterone with or without the use of GnRH agonist downregulation. The correct duration for exposure to progesterone is still not well established. To date, there are no prospective randomized trials available, comparing different durations of progesterone supplementation before the date of transfer, with regard to treatment outcome (Nawroth).

In this trial, the investigators want to determine the optimal duration of progesterone supplementation: 3 or 5 days before embryo transfer.

DETAILED DESCRIPTION:
The purpose is to transfer the embryo during the 'window of implantation', what is defined as the period during which the uterus is receptive for implantation of the free-lying blastocyst. This has been a subject of debate since many years (Bourgain et al, 2007).

Succesful implantation requires a co-ordinated series of events allowing a timely dialogue between a receptive endometrium and the intrusive blastocyst (Tabibzadeh, 1998). The period of receptivity is thought to be 3 days in human (Rogers et al, 1989; Yoshinaga, 1988; Psychoyos, 1993; Harper, 1992). It is suggested that blastocyst apposition begins about day LH+6 and is completed by day LH+10 (Lessey, 2000).

A number of structural and functional endometrial changes have been suggested to play a role in the implantation process: the formation of luminal epithelial pinopodes (Enders et al, 1973), expression of adhesion molecules and growth factors and cytokines (Lessey, 2000). Most of them are related directly or indirectly to progesterone secretion and influence on the endometrium.

In the Centre of Reproductive Medicine of the Brussels University Hospital, the investigators start progesterone supplementation 5 days before the transfer of a day 3 embryo. In order to mimic the natural cycle, since progesterone starts to rise 2 to 3 days before ovulation, due to the LH-stimulated production by the peripheral granulosa cells (Speroff). In fresh IVF-cycles, progesterone is started from the day of oocyte retrieval. HCG administration in fresh cycles will lead to an increase in progesterone levels and therefore, endometrium will progress quickly, compared with frozen-thawed cycles which are hormone supplemented (Nawroth).

In other centres, progesterone supplementation is generally started 3 days before the embryo transfer.

In this trial, the investigators want to determine the optimal duration of progesterone supplementation: 3 or 5 days before embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* Artificial cycles, in which a frozen-thawed day 3 embryo is replaced.
* Signed informed consent.
* Normal transvaginal ultrasound at screening, without evidence of clinically significant abnormality consistent with finding adequate for ART with respect to uterus and adnexa.
* Embryos must be frozen by vitrification technique (cfr supra).
* Single or dual embryo transfer.
* Recipients of oocyte donation cycles may be included.

Exclusion Criteria:

* Known allergic reactions to progesterone products.
* Intake of experimental drug within 30 days prior to study start.
* Contraindication for pregnancy.
* Embryos of women above 39 years of age at the time of embryo freezing.

Max Age: 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2012-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate | 7 weeks of pregnancy

SECONDARY OUTCOMES:
live birth rate | 9 months after embryo transfer

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Belgium

REFERENCES:
- [Derived] van de Vijver A, Polyzos NP, Van Landuyt L, Mackens S, Stoop D, Camus M, De Vos M, Tournaye H, Blockeel C. What is the optimal duration of progesterone administration before transferring a vitrified-warmed cleavage stage embryo? A randomized controlled trial. Hum Reprod. 2016 May;31(5):1097-104. doi: 10.1093/humrep/dew045. Epub 2016 Mar 22. PMID 27005893